CLINICAL TRIAL: NCT03581591
Title: An Open Label Trial to Assess the Safety and Efficacy of Burosumab (KRN23), an Investigational Antibody to FGF23, in a Single Pediatric Patient With Epidermal Nevus Syndrome(ENS) and Associated Hypophosphatemic Rickets
Brief Title: Open Label Trial Assessing Safety and Efficacy of Burosumab (KRN23), in a Patient With ENS and Hypophosphatemic Rickets
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Redwood Dermatology Sciences (Other)
Collaborators: Ultragenyx Pharmaceutical Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ENSKRN23.1
Record Dates: First submitted 2017-10-27; First posted 2018-07-10 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Hypophosphatemia; Hypophosphatemic Rickets; Pain, Chronic
MeSH Terms: conditions — Hypophosphatemia; Rickets, Hypophosphatemic; Chronic Pain | interventions — burosumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Primary; open label (Experimental): Injection of Burosumab every two to three weeks based on Serum Phosphorus level of subject. Initial dose to be 0.3 mg/kg. Subsequent dosing will be titrated up or down depending on Serum Phosphorus level for that time period.
  Interventions: Biological: Burosumab

INTERVENTIONS:
Biological: Burosumab — recombinant human IgG1 monoclonal antibody to fibroblast growth factor 23)

SUMMARY:
A 52 week, open label trial to assess the safety and efficacy of KRN23, an investigational antibody to FGF23, in a single pediatric patient with Epidermal Nevus Syndrome(ENS) and associated hypophosphatemic rickets

A 26 weeks extension to original study to monitor patient lab results for her safety.

DETAILED DESCRIPTION:
1.1 Primary Objective

The effect of KRN23 treatment on normalizing age-adjusted serum phosphorous levels in a single pediatric patient with Epidermal Nevus Syndrome associated hypophosphatemic rickets

1.2 Secondary Objectives

1. The PD profile of KRN23 as assessed by changes from baseline over time 1,25(OH)2D, iPTH, Serum Calcium, TRP and TmP/GFR (the ratio of renal tubular maximum phosphate reabsorption rate to glomerular filtration rate)
2. Changes in underlying skeletal disease/rickets as assessed by standard radiographs utilizing the Radiographic Global Impression of Change (RGI-C) rating scales
3. Effects of KRN23 on biochemical markers of bone turnover that reflect rickets severity, alkaline phosphatase (ALP)
4. Walking ability as assessed by 6-Minute Walk Test (6MWT)
5. Patient/parent-Reported Outcomes as assessed by PROMIS and FPS-R rating scales

1.3 Exploratory Objective

1. Dual-energy X-ray absorptiometry (DXA)

1.4 Safety Objective Assess the safety of KRN23 administration in a single patient with ENS-associated hypophosphatemic rickets, based on adverse events (AEs), laboratory assessments, cardiac imaging and renal ultrasound.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has confirmed ENS by physician diagnosis
2. Patient has confirmed FGF23 elevations in the context of low serum phosphorous < 4.1 mg/dL
3. Patient able to tolerate KRN23 treatment
4. Have a corrected serum calcium level < 10.8mg/dL
5. Have an eGFR >60 ml/min
6. Must be willing in the opinion of the investigator, to comply with study procedures and schedule
7. Provide written informed consent by a parent after the study has been explained and prior to any research related procedures begin

Exclusion Criteria:

1. Concomitant use of active vitamin D (i.e calcitriol) and/or exogenous phosphate supplementation. Patient will be allowed OTC Vitamin D should levels drop below <20 ng/ml
2. The use or enrollment in studies using other investigational therapies including other monoclonal antibodies
3. Subject and their parent not willing or not able to give written informed consent
4. In the Investigators opinion, the patient may not be able to meet all the requirements for study participation
5. Patient has a history of hypersensitivity to KRN23 excipients that in the opinion of the investigator, places the patient at an increased risk of adverse effects
6. Patient has a condition that in the opinion of the investigator could present a concern for subject safety or data interpretation.

Max Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1 (Actual)
Dates: Start 2018-01-31 (Actual); Primary Completion 2019-12-06 (Actual); Study Completion 2019-12-06 (Actual)

PRIMARY OUTCOMES:
The effect of KRN23 treatment on normalizing age-adjusted serum phosphorous levels in a single pediatric patient with Epidermal Nevus Syndrome associated hypophosphatemic rickets | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Sugarman, MD PhD, Principal Investigator — Redwood Dermatology Sciences
Locations (1):
- The Focus Center, PC, Clinton, Utah, United States

REFERENCES:
- [Background] Aono Y, Yamazaki Y, Yasutake J, Kawata T, Hasegawa H, Urakawa I, Fujita T, Wada M, Yamashita T, Fukumoto S, Shimada T. Therapeutic effects of anti-FGF23 antibodies in hypophosphatemic rickets/osteomalacia. J Bone Miner Res. 2009 Nov;24(11):1879-88. doi: 10.1359/jbmr.090509. PMID 19419316
- [Background] Aono Y, Hasegawa H, Yamazaki Y, Shimada T, Fujita T, Yamashita T, Fukumoto S. Anti-FGF-23 neutralizing antibodies ameliorate muscle weakness and decreased spontaneous movement of Hyp mice. J Bone Miner Res. 2011 Apr;26(4):803-10. doi: 10.1002/jbmr.275. PMID 20939065
- [Background] Carpenter TO, Imel EA, Ruppe MD, Weber TJ, Klausner MA, Wooddell MM, Kawakami T, Ito T, Zhang X, Humphrey J, Insogna KL, Peacock M. Randomized trial of the anti-FGF23 antibody KRN23 in X-linked hypophosphatemia. J Clin Invest. 2014 Apr;124(4):1587-97. doi: 10.1172/JCI72829. Epub 2014 Feb 24. PMID 24569459
- [Background] Lim YH, Ovejero D, Sugarman JS, Deklotz CM, Maruri A, Eichenfield LF, Kelley PK, Juppner H, Gottschalk M, Tifft CJ, Gafni RI, Boyce AM, Cowen EW, Bhattacharyya N, Guthrie LC, Gahl WA, Golas G, Loring EC, Overton JD, Mane SM, Lifton RP, Levy ML, Collins MT, Choate KA. Multilineage somatic activating mutations in HRAS and NRAS cause mosaic cutaneous and skeletal lesions, elevated FGF23 and hypophosphatemia. Hum Mol Genet. 2014 Jan 15;23(2):397-407. doi: 10.1093/hmg/ddt429. Epub 2013 Sep 4. PMID 24006476